CLINICAL TRIAL: NCT03461926
Title: Using a Combined Health Action Process Approach and mHealth Intervention to Increase Non-Sedentary Behaviours in Office-Working Adults - A Randomized Controlled Trial
Brief Title: A Combined HAPA and mHealth Intervention to Increase Non-Sedentary Behaviours in Office-Working Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Dr. Harry Prapavessis, Professor, Western University, Canada
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: HAPA Planning and SB in OWA
Record Dates: First submitted 2018-02-26; First posted 2018-03-12 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Sedentary Lifestyle; Health Behaviour Change
Keywords: Sedentary Behaviour; Health Behaviour Change; Health Action Process Approach; mHealth; Intervention; Non-Sedentary Behaviours; Break Frequency; Break Duration; Action Planning; Coping Planning; Work Performance; Health Outcomes
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: This study will employ a prospective, 2-group, repeated measure (2x5), randomized controlled trial design. All participants will be randomized into either a 6-week HAPA-treatment (SB-related planning + text messages intervention) or waitlisted control (no treatment) condition. All primary outcomes will be assessed at four time points (baseline, 2, 4, and 6 weeks), and again at a two-week follow-up (8 weeks). Action and coping planning and action control towards reducing workplace sitting time will be assessed at the same time points. Secondary outcome assessments (i.e., work- and health-related outcomes) will occur pre- (baseline) and post-intervention (6 weeks).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HAPA-treatment (Experimental): (SB-related planning + daily text messages)
  Interventions: Behavioral: (SB-related planning + daily text messages)
- Control (No Intervention): (No Treatment) Participants randomly assigned to the control group will receive no information or intervention of any kind and will only be asked to complete the outcome questionnaires.

INTERVENTIONS:
Behavioral: (SB-related planning + daily text messages) — Participants will receive a one-on-one behavioral counseling session, and planning sheet as reference for developing strategies as part of their Action/Coping Plan. Participants will be asked to form 3-4 actions/coping plans specifying when, where, how, and for how long they would reduce workplace sitting time; and anticipate potential barriers and identify ways they could be overcome. Strategies will focus on increasing break frequency to every 30-45 minutes, achieving a break duration of 2-3 minutes, and increasing standing and light-intensity PA time, during work hours. Participants will receive sedentary behaviour-related text messages twice daily, depending on their preferences and schedule, which will act as mini-booster interventions.
  Arms: HAPA-treatment

SUMMARY:
Societal changes have resulted in reduced demands to be active and increased daily time spent sitting. Sedentary behavior (SB) has been linked to many health problems such as type 2 diabetes and heart disease. Office-working adults are a high-risk population for excessive SB. Increasing the length and frequency of breaks from sitting and increasing the time spent standing and engaged in light physical activity are ways to decrease SB. The purpose of this study is to determine whether combining a Health Action Process Approach-based (theory-driven), specifically action and coping planning intervention, with a tailored text messaging intervention can reduce workplace sitting time among adult office workers. Participants in the intervention group will receive one behavioural counselling session, followed by daily, tailored text messages over a 6-week period, with a focus on encouraging them to reduce their occupational sitting time by increasing their frequency and duration of breaks from sitting, as well as time spent standing and engaged in light-intensity physical activity. It is expected that office-working adults who receive the planning intervention and tailored text messages will report greater increases in non-sedentary behaviours (e.g., break frequency, break duration, standing, light physical activity) than those who do not receive the intervention.

DETAILED DESCRIPTION:
Using a randomized controlled trial design, the purpose of this study will be to examine whether combining a HAPA-based intervention, specifically action and coping planning, with a tailored text message intervention can reduce workplace sitting time by increasing frequency and length of breaks from sitting and non-exercise activity thermogenesis (NEAT) behaviours (i.e., standing, light-intensity physical activity) among office-working adults. A secondary purpose will be to examine the effects of the intervention on participants' action planning, coping planning and action control regarding reducing their workplace sitting time, as well as self-rated work performance and health-related outcomes (i.e., role limitations due to physical health, role limitations due to personal or emotional problems, emotional well-being, and energy/fatigue). Another secondary objective will be to determine if action and coping planning and action control towards reducing workplace sitting time are related to actual break behaviour, time spent standing, and time spent in light-intensity physical activity.

If successful, participants in the intervention group (sedentary intervention group) will report reduced workplace sitting time, and greater break frequency and break duration, time spent standing, and time spent in light-intensity physical activity, compared to participants in the control group (no treatment). In addition, it is hypothesized that participants in the intervention group will report greater action and coping planning and action control towards reducing workplace sitting time, as well as improved work- and health-related outcomes.

This study will employ a prospective, 2-group, repeated measures, randomized controlled trial (RCT) design. Participants will be full-time adult, office workers primarily recruited from large businesses and office spaces.

Potential participants (estimated enrolment: 112) will be recruited by Andrew Scott Rollo, Principal Investigator, for this study. Relevant contacts/liaisons and/or senior executives (i.e., Head of Human Resources, President, Chief Executive Officer, Office Manager) at potential businesses of interest will be sought out via publically available sources (e.g., London Chamber of Commerce Business Directory, company websites, etc.) and contacted via email. The email will include a letter of information (LOI) and recruitment poster and request the individual's assistance with recruitment. For each business/office, if the individual accepts the invitation and informs the researchers that he/she is willing to aid with the recruitment process, the individual will then be asked to email all full-time employees in their respective office/business and offer them the opportunity to participate. In this recruitment email, the recruitment poster and Letter of Information will be provided. Participants will be instructed to contact the researcher via email and/or phone if they wish to participate or receive additional details prior to making a decision as to whether to participate. A second recruitment approach will involve recruiting full-time adult, office workers through recruitment posters distributed through social media (i.e., Facebook, LinkedIn) and public advertisements (i.e., transit stations, newspapers). The study will also be advertised through emails sent out to various faculties at Western University. Recruitment posters and LOIs will be posted on social media and in public spaces. As stated previous, office-workers interested in the study will be instructed to contact the researcher via email and/or phone to sign up for study participation.

At this point of contact, an email response will be sent to any interested individual. Adult office-workers who choose to take part in this study will receive a link via email that directs them to the Letter of Information, Informed Consent, and questionnaire for assessment of baseline measurements, which will be administered through a third party website called SoSci (online survey service). Participants will be assured that participation in this study is voluntary, that they are free to discontinue and withdraw from the study at any time, and that they may choose to skip any questions that they do not wish to answer without any effect on their employment status/work conditions. In other words, refusing to participate, refusing to answer any questions or withdrawing from the study will not impact their employment beyond potentially not receiving benefits associated with study participation. After viewing the Letter of Information and indicating that they consent to participate in the study (by clicking "I agree" on the survey), participants will be asked to complete a brief demographics questionnaire, followed by a questionnaire for baseline assessment of primary and secondary outcomes. In the initial email response sent to potential participants, participants randomized into the intervention group will also be asked to provide a day and time (within 3 days of completing the baseline assessment) that they would be available to schedule the behavioural counselling session they will receive.

Upon completion of the Baseline assessment and prior to intervention delivery, all participants will be randomized, using computer-generated randomized stratification, into either a 6-week HAPA-treatment (SB-related planning + text messages intervention) or waitlisted control (no treatment) condition. For those in the treatment group, the study objective will be to reduce workplace sitting time by increasing non-sedentary or NEAT behaviours (i.e., increasing break frequency to a break every 30-45 minutes, with each break having a duration of 2-4 minutes, and increasing their time spent standing and engaged in light-intensity PA. Participants randomly assigned to the control group will receive no information or intervention of any kind and will only be asked to complete the outcome questionnaires.

At the agreed upon and scheduled time, the researcher will deliver the intervention (i.e., implement the appropriate HAPA-based behavioural counselling session involving action and coping planning) either in person OR electronically via phone and an online presentation website (www.zoho.com). The method of delivery will entirely depend on the participant's availability, preference, and whether they live within driving distance of the investigator. To ensure equal numbers of local and remote participants in both conditions, two computer-generated random number lists will be created by the lead investigator using an online research randomization program. Participants will be asked to complete a second informed consent (written informed consent) at this time.

The one-on-one counseling sessions will be delivered by the principal investigator to ensure standardization between participants. During the counseling session, the researcher will first ask if the participant has any strategies that he/she would like to try or think would be effective. As much as possible, strategies will be kept as original and specific to the participant's lifestyle as possible, while still fulfilling the study objectives. Upon creation of each strategy, the researcher will ask the participant if they think that the strategy they came up with is realistic. The number of strategies will also be personalized depending on how the participant's baseline measures compare to the objectives of their treatment group. This will be done in order to attenuate for any neglected/unused strategies by those with larger differences between baseline and objective values. Similarly, coping strategies will be created alongside each strategy in order to boost the adherence to the developed strategies. When an action plan strategy is developed, the researcher will ask the participant "what are some challenges you foresee with executing this strategy?", followed by "what do you think is something we can do in order to overcome this/these challenges?" This will be done in order to keep the coping strategies personalized to the participant's lifestyle. Overall, the behavioral counseling sessions will take between 20-30 minutes to complete and both groups will receive equal contact time. Participants will be given the form with their action plan and coping strategies and told to display it somewhere prominent so they will be reminded of the strategies. The principal investigator will conduct the planning interventions in a non-interfering manner by providing brief instructions and then remaining available to answer any questions.

At this point, participants in the intervention group will then be entered into a contact list on the text-messaging website called "Oh Don't Forget." "Oh Don't Forget," is a Web-based application that works through "Recess Mobile" to send messages from a computer to mobile phone numbers that are programmed into the application. All participants will begin receiving tailored text messages the day after receiving their one-on-one counseling session. Every participant will receive the same daily texts as each other participant in their group, with times varying slightly depending on their schedule. As planning is an ongoing process, participants will be reminded (via text message) to formulate another set of action and coping plans at the beginning of weeks 3 and 5. Upon completion of the intervention period at 6 weeks, participants will be notified that they will no longer be receiving text messages and that the study is completed.

After the initial behavioural counseling session, participants will be told they will receive a link to a questionnaire (assessment of primary and secondary outcomes) in their email every 2 weeks, for the next 6 weeks (i.e., weeks 2, 4, and 6), and to complete the questionnaire the day they receive it. Participants will also be told that 2 weeks following the end of the 6-week intervention, there will be a follow-up questionnaire (week 8), which they will receive and be asked to complete. All primary and secondary outcome questionnaires will be completed online and administered through a third party website called SoSci (online survey service). Participants will also be reminded via text to complete these. Primary outcomes including frequency of breaks, length of breaks, and NEAT behaviours at work (i.e., standing, light-intensity PA) will be assessed using subjective, self-report approaches. Secondary analyses will be performed to examine effects of the intervention on theoretical determinants of behaviour change (i.e., action planning, coping planning, action control), as well as participants' perceived work-related outcomes (i.e., self-rated work performance) and health-related outcomes (i.e., role limitations due to physical health, role limitations due to personal or emotional problems, emotional well-being, and energy/fatigue). All primary outcomes will be assessed at four time points (baseline, 2, 4, and 6 weeks), and again at a two-week follow-up (8 weeks). Action and coping planning and action control towards reducing workplace sitting time will be assessed at the same time points. Secondary outcome variables (i.e., perceived work- and health-related outcomes) will be assessed pre- (baseline) and post-intervention (6 weeks).

ELIGIBILITY:
Inclusion Criteria:

* To be eligible to participate, participants must: (a) be 18+ years of age, (b) be a full-time worker/employee in an office setting, (c) be in self-reported good mental and physical health, (d) be able to read and write in English, (e) have access to a computer with Internet, and (f) own a mobile phone with free unlimited incoming text messages.

Exclusion Criteria:

* Individuals who are under 18 years of age, do not read or write in English, are not full-time workers/employees in office settings, do not have access to a computer with Internet, and/or do not own a mobile phone with free unlimited incoming text messages and/or emails are not eligible to participate in this study. Additional exclusion criteria include any individual who is pregnant and/or suffering from a medical condition that prohibits them from being physically active.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Changes in Frequency of Breaks from Sitting at Work | Baseline, Weeks 2, 4, 6, and at the 2-week follow-up (Week 8)
  Modified version of the SIT-Q 7d (Wijndaele et al., 2014; Sui & Prapavessis, 2016); 1-item; 12-point scale
Changes in Duration of Breaks from Sitting at Work | Baseline, Weeks 2, 4, 6, and at the 2-week follow-up (Week 8)
  Modified version of the SIT-Q 7d (Wijndaele et al., 2014; Sui & Prapavessis, 2016); 1-item; 10-point scale
Changes in Time Spent Standing at Work | Baseline, Weeks 2, 4, 6, and at the 2-week follow-up (Week 8)
  Five-item modified Occupational Sitting and Physical Activity Questionnaire (OSPAQ; Chau, Van Der Ploeg, Dunn, Kurko, & Bauman, 2012)
Changes in Time Spent Engaged in Light-Intensity Physical Activity (i.e., walking) at Work | Baseline, Weeks 2, 4, 6, and at the 2-week follow-up (Week 8)
  Five-item modified Occupational Sitting and Physical Activity Questionnaire (OSPAQ; Chau, Van Der Ploeg, Dunn, Kurko, & Bauman, 2012)
Changes in Time Spent Sitting at Work | Baseline, Weeks 2, 4, 6, and at the 2-week follow-up (Week 8)
  Five-item modified Occupational Sitting and Physical Activity Questionnaire (OSPAQ; Chau, Van Der Ploeg, Dunn, Kurko, & Bauman, 2012); value: Minutes/Day

SECONDARY OUTCOMES:
Action Planning towards reducing workplace sitting time | Baseline, Weeks 2, 4, 6, and at the 2-week follow-up (Week 8)
  Four-items; five-point Likert scale (1 = "completely disagree" to 5 = "totally agree")
Coping Planning towards reducing workplace sitting time | Baseline, Weeks 2, 4, 6, and at the 2-week follow-up (Week 8)
  Five-items; five-point Likert scale (1 = "completely disagree" to 5 = "totally agree")
Action Control towards reducing workplace sitting time | Baseline, Weeks 2, 4, 6, and at the 2-week follow-up (Week 8)
  Six-items; five-point Likert scale (1 = "completely disagree" to 5 = "totally agree")
Self-rated Work Performance | Baseline, Week 6
  One-item, 11-point Likert scale
Role limitations due to physical health | Baseline, Week 6
  RAND 36-item Short Form Survey (SF-36; Ware and Sherbourne, 1992) modified version (16-item). Four-items will assess participant's perceived role limitations due to physical health problems; 2-point scale (yes, no)
Role limitations due to emotional health | Baseline, Week 6
  RAND 36-item Short Form Survey (SF-36; Ware and Sherbourne, 1992) modified version (16-item). Three-items will assess role limitations due to personal or emotional problems; 2-point scale (yes, no)
Emotional well-being | Baseline, Week 6
  RAND 36-item Short Form Survey (SF-36; Ware and Sherbourne, 1992) modified version (16-item). Five-items will assess perceived emotional well-being; 5-point Likert scale (All of the time =1, Most of the time = 2, Some of the time = 3, A little of the time = 4, None of the time = 5)
Energy/Fatigue | Baseline, Week 6
  RAND 36-item Short Form Survey (SF-36; Ware and Sherbourne, 1992) modified version (16-item). Four-items will assess perceived energy/fatigue; 5-point Likert scale (All of the time =1, Most of the time = 2, Some of the time = 3, A little of the time = 4, None of the time = 5)

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Western Ontario, London, Ontario, Canada

REFERENCES:
- [Derived] Rollo S, Prapavessis H. A Combined Health Action Process Approach and mHealth Intervention to Increase Non-Sedentary Behaviours in Office-Working Adults-A Randomised Controlled Trial. Appl Psychol Health Well Being. 2020 Nov;12(3):660-686. doi: 10.1111/aphw.12201. Epub 2020 Apr 28. PMID 32342662